CLINICAL TRIAL: NCT06885515
Title: Short Telomeres in Familial and Sporadic Fibrotic Interstitial Lung Diseases in Israel
Brief Title: Telomeres Length in Israeli Fibrotic ILD Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Barzilai Medical Center (Other)
Collaborators: Tel Aviv Medical Center (Other); Israel Society of Pulmonology (Unknown)
Responsible Party: Principal Investigator, Dr. Ori Wand, Head, Division of Pulmonary Medicine, Barzilai Medical Center
Other Study IDs: BRZ-0050-24
Record Dates: First submitted 2025-03-09; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Fibrosis
Keywords: pulmonary fibrosis; familial interstitial lung disease; familial pulmonary fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- familial pulmonary fibrosis: Patients with familial pulmonary fibrosis are those with at-least one first-degree or second-degree relative with FILD
  Interventions: Diagnostic Test: leukocyte telomere length (LTL) will be measured using the Telomere Restriction Fragment (TRF) Analysis method
- non familial pulmonary fibrosis: Patients with pulmonary fibrosis without relatives with FILD
  Interventions: Diagnostic Test: leukocyte telomere length (LTL) will be measured using the Telomere Restriction Fragment (TRF) Analysis method
- control: 10 healthy age-matched controls with no personal or family history of lung disease will be recruited as well
  Interventions: Diagnostic Test: leukocyte telomere length (LTL) will be measured using the Telomere Restriction Fragment (TRF) Analysis method

INTERVENTIONS:
Diagnostic Test: leukocyte telomere length (LTL) will be measured using the Telomere Restriction Fragment (TRF) Analysis method — genomic DNA (2-5 µg) is digested overnight at 37°C with HinfI restriction endonuclease. Fragments are being separated on an agarose gel, transferred to a Hybond N+ membrane. The membrane is being hybridized over night at 50°C with a 5' end-labeled (AACCCT)3 oligonucleotide probe and with ladder probe of 1Kb ladder. Following membrane washes the membrane is exposed to PhosphoImager. The mean telomere length is calculated by the computer program Telotool [19-20]. TRF analysis will be conducted at the laboratory of Prof. Yehuda Tzfati at the Hebrew University, which is highly experienced in the field of telomere biology and in telomere length analysis. Blood samples will be taken once from each participant. no genetic sequencing will be performed as part of this study.

SUMMARY:
Individuals with fibrotic interstitial lung diseases (FILD) will be recruited after providing informed consent. in addition to routine data as usually collected in the clinic, blood samples will be taken for measurement of telomeres length in peripheral blood leukocytes using the Telomere Restriction Fragment (TRF) Analysis method. Participants with FILD will be followed-up for 1-year after recruitment, including clinical and pulmonary function tests at-least every 6 months, or more frequently, according to the treating physician discretion.

DETAILED DESCRIPTION:
Scientific Background Interstitial lung diseases (ILD) comprise a large heterogenic group of conditions which involve the lung parenchyma by inflammation, fibrosis, or both. Fibrotic ILD (FILD), which are characterized by evidence of lung fibrosis by either imaging studies (chest CT), and/or histopathology, may result from known exposures or association, or be idiopathic. Management of FILD depends on specific diagnosis, patient characteristics, and disease behavior. Some conditions may respond favorably to immunosuppression, while in others, such as idiopathic pulmonary fibrosis (IPF), such treatment may be harmful. Antifibrotic therapy may attenuate the progression of various FILD, including IPF, yet in many cases, disease progression ultimately leads to a fatal outcome or need for lung transplantation.

Telomeres are repetitive 6-nucleotide sequences which cap the end of chromosomes, and are essential in stabilizing chromosomes [1]. While they shorten with each cell replication, telomeres are maintained by complex mechanisms which can add nucleotide repeats (telomerase), and protect chromosomal ends by other mechanisms. Shortened telomeres may result from mutations in telomere related genes. Short telomeres have also been associated with single nucleotide polymorphism in those genes. Telomeres shorten with age, and are also shorter among males. Additional acquired factors also contribute to shortening, including harmful exposures, cigarette smoking, obesity, stress, lack of physical activity, and others [3-4].

Short leukocyte telomere length (LTL), i.e. <10th percentile adjusted for age, are common in patients with various FILD, with or without identifiable mutations in telomere related genes, both in familial and sporadic cases [5-6]. Short LTL has been associated with worse prognosis among subjects with several FILD, including faster deterioration of pulmonary functions tests, quicker disease progression, and shorter transplant-free survival [7-11]. In addition, IPF patients with short LTL had worse prognosis when exposed to immunosuppressive treatment [12], as were patients with other FILD commonly treated with immunosuppression [13]. Antifibrotic therapy, on the other hand, seems to be safe and effective [14].

This accumulating data has implications on the management of patients. Experts suggest testing for LTL in patients with familial pulmonary fibrosis, early age of disease onset, or with personal or family history of relevant extrapulmonary disease [8, 15]. Prompt initiation of antifibrotics, early referral for lung transplant and avoidance of immunosuppression have also been recommended [8, 16].

However, the prevalence of short LTL varies among ethnically diverse cohorts of FILD patients [7] and have never been assessed in the Israeli population.

Rationale We believe that this study will shed light on the prevalence of short LTL in Israeli individuals with FILD, and identify predictors which will enable more precise targeting of LTL measurements in Israel. In addition, it may guide physicians with regards to careful administration of immunosuppressive treatments in Israeli FILD patients suspected of having short telomeres.

Hypothesis We believe that the proportion of subjects with short LTL is higher in Israeli subjects with familial FILD than with sporadic FILD, yet that a significant proportion of sporadic FILD subjects will also have short LTL.

This may lead to more widespread and evidence-based directed use of LTL measurements among Israeli patients with FILD.

Study Objectives General Aim To assess the prevalence of short LTL among Israeli patients with FILD, and identify relevant association and impact of short LTL on those patients.

Specific Aims

1. To assess the prevalence of short LTL among Israeli patients with familial and sporadic FILD.
2. To identify risk factors for short LTL in Israeli FILD patients.
3. To prospectively assess the outcome of participants (with and without short telomeres) using a composite of death of any cause, lung transplantation, and forced vital capacity (FVC) decline ≥5% over a 1-year period [17].
4. Additionally, we will conduct an exploratory analysis of the components of the composite outcome measure as well as other possible criteria for progressive pulmonary fibrosis (PPF), including annual decline of diffusion capacity for CO (DLCO) ≥10%, FVC decline ≥10%, FVC decline 5-9%, DLCO decline ≥15%, CT progression of fibrosis, and clinical worsening of symptoms [17, 18].

Research Design & Methods This is a prospective study, with collaboration of two Medical Centers: The Pulmonary Fibrosis Center of Tel-Aviv Medical Center (Ichilov), a tertiary medical center in Central Israel, and the Division of Pulmonary Medicine of Barzilai University Medical Center, a secondary, peripheral medical center from Southern Israel.

A total of 90 patients with FILD will be recruited from the two clinics, thus representing diverse Israeli population. This cohort will include 30 patients with familial pulmonary fibrosis and 60 with sporadic lung fibrosis.

Patients with familial pulmonary fibrosis are those with at-least one first-degree or second-degree relative with FILD [8].

10 healthy age-matched controls with no personal or family history of lung disease will be recruited as well.

Thus, sample size of the whole study, as well as in our Center will include up to 100 participants.

Participants with FILD will be followed-up for 1-year after recruitment, including clinical and pulmonary function tests at-least every 6 months, or more frequently, according to the treating physician discretion. Collected data will include participants' demographics and anthropometrics, family history and personal medical history, pulmonary function tests results, thoracic imaging and histopathological patterns, clinical diagnoses of FILD (according to a multidisciplinary team discussion), treatment and outcome.

Measured Variables

Collected data will include (see attached excel file data sheet):

* Age
* Gender
* Ethnic group
* Birthplace
* Height, weight, BMI
* Family history
* Smoking history
* Place of residence
* Occupation
* Past medical history, co-morbidities, and medications
* Relevant exposures
* ILD diagnosis
* Specific ILD therapies
* Clinical findings, including physical examination, laboratory tests, pulmonary function tests, imaging, echocardiography, lung biopsy diagnosis, bronchoalveolar lavage differential
* Hospitalizations
* Diagnosis of lung cancer or other malignancy
* Outcomes, including annual decline of pulmonary function tests, worsening symptoms, worsening CT signs of lung fibrosis, lung transplantation, and death

LTL measurement In addition to clinical data, blood samples will be collected to measure LTL using the "gold standard" Telomere Restriction Fragment (TRF) Analysis method. In short, genomic DNA (2-5 µg) is digested overnight at 37°C with HinfI restriction endonuclease. Fragments are being separated on an agarose gel, transferred to a Hybond N+ membrane. The membrane is being hybridized over night at 50°C with a 5' end-labeled (AACCCT)3 oligonucleotide probe and with ladder probe of 1Kb ladder. Following membrane washes the membrane is exposed to PhosphoImager. The mean telomere length is calculated by the computer program Telotool [19-20]. TRF analysis will be conducted at the laboratory of Prof. Yehuda Tzfati at the Hebrew University, which is highly experienced in the field of telomere biology and in telomere length analysis. Blood samples will be taken once from each participant. As detailed above for LTL measuremement, no genetic sequencing will be performed as part of this study.

Sample Size Calculation Assuming that 50% and 20% of participants in the familial FILD and sporadic FILD will have short LTL, a sample size of 87 patients (29 familial and 58 sporadic FILD) is required to detect significant differences in the proportions of subjects with short LTL with an alpha error rate of 0.05 and 80% power.

The proposed study will require approval by local Institutional Review Boards and Helsinki Committees of both Medical Center. Individuals will provide informed consent prior to participation in the study.

Inclusion Criteria

1. Adult subjects, aged ≥18-years-old
2. Able and willing to provide informed consent to participate in the study
3. Lung fibrosis evident on chest CT (signs of honeycombing and/or traction bronchiectasis) [17]
4. Subjects fulfilling criteria 1 and 2 but with no evidence of chronic lung disease will serve as controls Exclusion Criteria

1. Subjects with sarcoidosis as the etiology for FILD 2. Subjects who had undergone lung transplantation 3. Pregnant women

Statistical Analysis Comparison between groups (i.e., familial vs sporadic FILD, patients with vs without short LTL) will be performed using Chi-square test, Mann-Whitney test, or Student's T-test, according to measured variables. Correlations will be assessed by calculating Pearson's or Spearman's coefficients, as appropriate. Assessing predictors of short LTL and of disease progression will be analyzed using univariate and multivariate logistic regression analysis models.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects, aged ≥18-years-old
2. Able and willing to provide informed consent to participate in the study
3. Lung fibrosis evident on chest CT (signs of honeycombing and/or traction bronchiectasis) [17]
4. Subjects fulfilling criteria 1 and 2 but with no evidence of chronic lung disease will serve as controls

Exclusion Criteria:

1. Subjects with sarcoidosis as the etiology for FILD
2. Subjects who had undergone lung transplantation
3. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 90 patients with FILD will be recruited . This cohort will include 30 patients with familial pulmonary fibrosis and 60 with sporadic lung fibrosis.
  Patients with familial pulmonary fibrosis are those with at-least one first-degree or second-degree relative with FILD. 10 healthy age-matched controls with no personal or family history of lung disease will be recruited as controls.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
the prevalence of short LTL among Israeli patients with familial and sporadic FILD. | 1 year
  the prevalence of short LTL among Israeli patients with familial and sporadic FILD.

SECONDARY OUTCOMES:
Composite prospective outcome | 1-year
  a composite of death of any cause, lung transplantation, and forced vital capacity (FVC) decline ≥5% over a 1-year period
lung transplantation | 1-year
forced vital capacity (FVC) decline ≥5% | 1 year
  decline of FVC 5% from baseline or more
criteria for progressive pulmonary fibrosis (PPF) | 1 year
  a composite outcome which includes: annual decline of diffusion capacity for CO (DLCO) ≥10%, FVC decline ≥10%, FVC decline 5-9%, DLCO decline ≥15%, CT progression of fibrosis and clinical worsening
All cause mortality | 1 year
  death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Ori Wand, Dr., Principal Investigator — Barzilai University Medical Canter

IPD SHARING:
Plan to Share IPD: Yes
baseline chracteristics, PFT, CT results, telomere length results
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: December 31 2027-December 31 2030
Access Criteria: after reasonable request from PI